CLINICAL TRIAL: NCT03829124
Title: Comparison of Propofol Combine Ketamine Anesthesia and Propofol Anesthesia in Schizophrenia Electroconvulsive Therapy: A Randomized Controlled Trial
Brief Title: Comparison of Ketamine Combine Propofol vs Propofol Anesthesia in Schizophrenia Electroconvulsive Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201800056A3
Record Dates: First submitted 2019-01-13; First posted 2019-02-04 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia
Keywords: Electroconvulsive therapy; ketamine
MeSH Terms: conditions — Schizophrenia | interventions — Propofol; Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ketamine + propofol group (Experimental): use ketamine + propofol for ECT induction
  Interventions: Drug: Propofol; Drug: Ketamine
- propofol group (Active Comparator): use propofol only for ECT induction
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol 10mg/ml IV push slowly 0.5-2mg/kg
Drug: Ketamine — Ketamine 50mg/ml IV push slowly 0.5- 1mg/kg
  Arms: ketamine + propofol group

SUMMARY:
Electroconvulsive therapy (ECT) serves as an effective adjuvant modality for major depressive disorder, schizophrenia, or bipolar affective disorder refractory to or contraindicated to psychopharmacological treatment. Anesthetics have been introduced into ECT sessions to alleviate ECT-inducing discomfort sensation, tachycardia, arrhythmia, hypertension, and anxiety.

Propofol is able to rapidly cross the blood-brain barrier (BBB), which leads to rapid onset of sedation and hypnosis. Meanwhile, propofol has hemodynamic depressant effect and attenuates hypertensive surge during ECT. Characteristics mentioned above make propofol one of widely used anesthetics for anesthetized ECT. However, propofol is also well known for anticonvulsant property. Thus, dosage of electrical stimulus may be increased to achieve ideal seizure quality in this setting, which also leads to higher risk of subsequent cognitive impairment or other complications.

Ketamine has also been widely used in the induction of anesthesia for the treatment of major depressive disease in recent years. It has been found to increase the permeability and therapeutic effect of antidepressants. Compared to traditional Barbiturate drugs or propofol, do not increase the threshold of electricity required by electroporation, which can reduce the time required for symptom relief of those drugs, It is a viable alternative induction drug.

There have been confirmed that ketamine combine propofol can be used for electroconvulsive treatment in patients with major depression and bipolar disorder, and even better Electroconvulsive quality can be obtained. Reduce the number of Electroconvulsive treatments and reduce the duration of treatment. However, the current literature has not yet verified the clinical benefit of ketamine combine propofol as an anesthetic induction drug in patients with schizophrenia who are receiving electroconvulsive therapy, and it is worthy of further study.

In the investigator's clinical practice, the purpose of this experiment is to explore: compared with propofol base anesthesia alone, and the combine use of ketamine and propofol may reduce the threshold of seizure, improve the quality of Electroconvulsive therapy and shorten the course of treatment. The combine use and titrate the drugs helps to reduce the side effects of both ketamine and propofol (such as cardiovascular side effects and positive symptoms) , achieve better Electroconvulsive therapy and effects.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) serves as an effective adjuvant or alternative modality for major depressive disorder, schizophrenia, or bipolar affective disorder refractory to or contraindicated to psychopharmacological treatment. Anesthetics have been introduced into ECT sessions to alleviate ECT-inducing discomfort sensation, tachycardia, arrhythmia, hypertension, and anxiety.

Propofol is highly lipid soluble and able to rapidly cross the blood-brain barrier (BBB), which leads to rapid onset of sedation and hypnosis. Meanwhile, propofol has hemodynamic depressant effect and attenuates hypertensive surge during ECT. Characteristics mentioned above make propofol one of widely used anesthetics for anesthetized ECT. However, propofol is also well known for anticonvulsant property, which may inevitably interfere with seizure propagation by electroconvulsive stimulus and diminish consequent efficacy. Thus, dosage of electrical stimulus may be increased to achieve ideal seizure quality in this setting, which also leads to higher risk of subsequent cognitive impairment or other complications.

Ketamine has also been widely used in the induction of anesthesia for the treatment of major depressive disease in recent years. It has been found to increase the permeability and therapeutic effect of antidepressants. Compared to traditional Barbiturate drugs or propofol, do not increase the threshold of electricity required by electroporation, which can reduce the time required for symptom relief of those drugs, It is a viable alternative induction drug. However, ketamine causes short-term dissociative symptoms, which may temporarily aggravate the positive symptoms of patients with schizophrenia after Electroconvulsive therapy, but the time of aggravation of positive symptoms generally does not exceed 30 minutes.

There have been many studies in the clinic, and it has been confirmed that ketamine combine propofol can be used for electroconvulsive treatment in patients with major depression and bipolar disorder, and even better Electroconvulsive quality can be obtained. Reduce the number of Electroconvulsive treatments and reduce the duration of treatment. However, the current literature has not yet verified the clinical benefit of ketamine combine propofol as an anesthetic induction drug in patients with schizophrenia who are receiving electroconvulsive therapy, and it is worthy of further study.

In the investigator's clinical practice, the purpose of this experiment is to explore: compared with propofol base anesthesia alone, and the combine use of ketamine and propofol may reduce the threshold of seizure, improve the quality of Electroconvulsive therapy and shorten the course of treatment. The combine use and titrate the drugs helps to reduce the side effects of both ketamine and propofol (such as cardiovascular side effects and positive symptoms) , achieve better Electroconvulsive therapy and effects.

ELIGIBILITY:
Inclusion Criteria:

* The clinical diagnosis is consistent with the schizophrenia, and the diagnostic requirements are in accordance with the Structural Diagnostic Interview Scale (SCID for Diagnostic and Statistical Manual of Mental Disorders (DSM-5)) and are recognized by psychiatrists as needing electroconvulsive therapy
* Vision and hearing that can be operated normally or corrected
* Subject consent form signed by the patient or agent

Exclusion Criteria:

* Past or recent diagnosis of neurocognitive impairment
* Contraindications for electroacupuncture treatment within one month, such as: myocardial infarction, cerebrovascular disease, Increase Intracranial pressure, cerebral hemangioma, untreated fracture, cervical spine injury, pheochromocytoma, heart failure, severe heart valve disease, deep Venous embolism, etc
* Untreated substances abuse disorder(eg illegal drugs, alcohol)
* Unspecified mental disorder
* PattientUnable to cooperate

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2019-05-24 (Estimated); Primary Completion 2021-01-19 (Estimated); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
The therapeutic effect after completing electroconvulsive treatment course | At baseline, after 3rd course treatment(average 1-2 week), after 6th course treatment(average 2-4 week), after completion of treatment course( average 4-6 weeks, up to 8 weeks)
  Record the change of disease illness, use The Clinical Global Impression - Improvement scale (CGI-I) and Clinical Global Impression - Severity scale (CGI-S) CGI-S(Severity) range 1-7 1: normal 7:extremely severe CGI-I(Improvement) range 1-7
  1:very much improved 7: vert much worse

SECONDARY OUTCOMES:
Change from baseline in Brief Psychiatric Rating Scale (BPRS) | At baseline, after 3rd course treatment(average 1-2 week), after 6th course treatment(average 2-4 week), after completion of treatment course( average 4-6 weeks, up to 8 weeks)
  Brief Psychiatric Rating Scale range:18-126
  Contains the following items:
  1. Somatic concern
  2. Anxiety
  3. Depression
  4. Suicidality
  5. Guilt
  6. Hostility
  7. Elated Mood
  8. Grandiosity
  9. Suspiciousness
  10. Hallucinations
  11. Unusual thought content
  12. Bizarre behaviour
  13. Self-neglect
  14. Disorientation
  15. Conceptual disorganisation
  16. Blunted affect
  17. Emotional withdrawal
  18. Motor retardation
  19. Tension
  20. Uncooperativeness
  21. Excitement
  22. Distractibility
  23. Motor hyperactivity
  24. Mannerisms and posturing Different item scores will have different results and outcomes
  ""Different values represent is not meaning a better or worse outcome, it must compare to the patient's status before""

IPD SHARING:
Plan to Share IPD: No